CLINICAL TRIAL: NCT06883084
Title: Clinical Relevance of the Pathologic Regression in Lymph Node for Locally Advanced Rectal Cancer Following Neoadjuvant Chemoradiotherapy: A Multi-center Study
Brief Title: Clinical Relevance of Pathologic Regression IN Lymph Node for Locally Advanced Rectal Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, M.D., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: GIH-SYSUSH14
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer; Lymph Node Metastasis
MeSH Terms: conditions — Rectal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We evaluated all related clinical and pathologic data of patients with Locally Advanced Rectal Cancer following Neoadjuvant Chemoradiotherapy, including the pathologic regression grading in the primary tumor site and lymph node, and other histopathologic characteristics. Finally, the present study was aimed at (1) clarifying the clinical significance of the Major Pathologic Regression for Locally Advanced Rectal Cancer following Locally Advanced Rectal Cancer in the primary tumor site and lymph node, and (2) comparing different Neoadjuvant Chemoradiotherapy treatments of this uncommon disease through conducting a large, multi-center cohort study.

DETAILED DESCRIPTION:
This large-scale, multi-center cohort study investigates the clinical significance of Pathologic Regression in lymph nodes (LNs) of patients with Locally Advanced Rectal Cancer (LARC) following Neoadjuvant Chemoradiotherapy (NCRT). Additionally, it compares the efficacy of diverse NCRT regimens in achieving pathologic regression and improving survival outcomes.

Study Design Type: Retrospective and prospective observational cohort study. Setting: Multi-center collaboration across 14 academic and community hospitals. Timeframe: Data from patients treated between 2014 and 2025 will be analyzed, with prospective follow-up ongoing until 2026.

Primary Objectives

Clarify the clinical significance of tumor regression in LN:

Define MPR thresholds for both primary tumor (e.g., ≤10% residual viable tumor) and lymph nodes (e.g., complete LN regression [ypN-Reg+] versus residual LN disease [ypN+]).

Correlate MPR status in the primary tumor and LNs with long-term outcomes:

Primary endpoints: Progression-Free Survival (PFS), Overall Survival (OS). Secondary endpoints: Local recurrence rate, distant metastasis-free survival.

Compare NCRT regimens:

Evaluate differences in MPR rates and survival outcomes between fluoropyrimidine-based, oxaliplatin-containing, and immunotherapy-augmented NCRT protocols.

Assess the impact of radiation dose escalation (e.g., 50.4 Gy vs. 45 Gy) on pathologic regression.

Study Population

Inclusion Criteria:

Adults (≥18 years) with histologically confirmed LARC (clinical stage II-III). Completion of NCRT followed by total mesorectal excision (TME). Availability of standardized pathologic reports and digitized whole-slide images (WSIs) for both primary tumor and LNs.

Exclusion Criteria:

Metastatic disease at diagnosis. Incomplete NCRT or surgical resection. Data Collection

Clinical Variables:

Demographics, NCRT regimen (drugs, doses, duration), surgical complications, adjuvant therapy, recurrence patterns.

Pathologic Variables:

Primary tumor: Residual viable tumor percentage, necrosis extent, tumor-infiltrating lymphocyte (TLS) density.

Lymph nodes: Regression grading (ypN-Reg+/-), number of regressed vs. metastatic LNs.

AI-driven quantitative analysis: Necrosis-to-tumor ratio (NECR-TD), TLS-to-necrosis ratio (T/NR), and spatial distribution of regressive features (Figure S2).

Imaging and Biomarkers:

Pre-treatment MRI-based tumor staging, post-treatment radiomic features (if available).

Statistical Analysis

Survival Analysis:

Kaplan-Meier curves and multivariable Cox regression to identify predictors of DFS/OS, adjusting for age, stage, and treatment regimen.

Subgroup analysis of LN regression (ypN-Reg+ vs. ypN-Reg-) in patients with ypN0 status.

Comparative Effectiveness:

Propensity score matching to balance baseline characteristics across NCRT regimens.

Meta-analysis of pooled multi-center data to assess heterogeneity in treatment effects.

Machine Learning:

Develop prognostic models integrating MPR status, histopathologic parameters, and clinical variables.

Ethical Considerations Approved by the Institutional Review Boards (IRBs) of all participating centers Innovation and Impact

Dual Focus on Primary Tumor and LNs:

First study to evaluate MPR thresholds simultaneously in primary tumor and LNs, addressing their independent prognostic roles.

Translational Insights:

Link LN regression to systemic immune responses (e.g., abscopal effect) and molecular heterogeneity between primary and metastatic sites.

Clinical Utility:

Provide evidence for standardizing MPR definitions in LARC and optimizing NCRT regimens based on tumor biology.

ELIGIBILITY:
Inclusion Criteria:

- Adults (≥18 years) diagnosed with locally advanced rectal adenocarcinoma (clinical stage II-III).

Completion of NCRT followed by curative-intent surgery. Availability of pre- and post-treatment histopathologic data, including standardized regression grading and digitized whole-slide images (WSIs).

Exclusion Criteria:

- distant Metastatic disease at diagnosis. Incomplete clinical or pathologic records.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Locally Advanced Rectal Cancer following Locally Advanced Rectal Cancer
Sampling Method: Probability Sample
Enrollment: 1080 (Estimated)
Dates: Start 2014-01-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
PFS | 10 years
  Progression free survival
OS | 10 years
  Overall survival